CLINICAL TRIAL: NCT05103371
Title: Examining the Feasibility and Effectiveness of a Prevention Program for Encouraging Self-care, Self-esteem, Body-esteem and Media Literacy Among Young Adolescents
Brief Title: A Prevention Program to Encourage Self-care, Self-esteem and Body-esteem Among Young Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tel Hai-Academic
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Primary Prevention
Keywords: prevention program; body-image; self-esteem; parents; adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Mili" prevention program, adolescents and active parents (Experimental): The program "Mili" will be delivered to adolescence aged 10-12, over 3 months. The program contains nine weekly, 90-min sessions that focus on Media literacy, self-esteem, self-image and body image. The parents will also participate by a phone app that will pass the parents activities to do with their children, in parallel to the program. All participants will complete a self-report questionnaire at baseline, after the program ends, and three months after the completion of the program.
  Interventions: Behavioral: Experiment: "Millie" prevention program, adolescents and active parents
- "Mili" prevention program, adolescents only (Active Comparator): The program "Mili" will be delivered to adolescence aged 10-12, over 3 months. The program contains nine weekly, 90-min sessions that focus on Media literacy, self-esteem, self-image and body image, no parental involvement in the program. Adolescents will complete a self-report questionnaire at baseline, after the program ends, and three months after the completion of the program.
  Interventions: Behavioral: Experiment: "Millie" prevention program, adolescents only
- control group (No Intervention): The control group will not receive the intervention program. The control group will complete the same self-report questionnaire as the intervention group at baseline, after the program ends, and three months after the completion of the program

INTERVENTIONS:
Behavioral: Experiment: "Millie" prevention program, adolescents and active parents — Prevention program: "Millie", with the participation of adolescents and parents
  Arms: "Mili" prevention program, adolescents and active parents
Behavioral: Experiment: "Millie" prevention program, adolescents only — Prevention program: "Millie", with the participation of adolescents only, no parental involvement in the program
  Arms: "Mili" prevention program, adolescents only

SUMMARY:
Cluster-Randomized Clinical trial, which includes the development and activation of an intervention program among young adolescents and their parents. Study hypothesis is that the intervention program will yield improvement in adolescents whose parents participated in the program, in comparison with the adolescents whose parents weren't involved in the intervention. Results will be measured using the study questionnaire, to be filled out by the participants before, after, and three months after the completion of the program. The questionnaire will include validated questionnaires with good psychometric qualities. The study protocol was approved by Tel Hai College institutional review board. Parents of all participants, in the intervention and in the control group, received information about the program and the study and were asked to provide informed consent.

DETAILED DESCRIPTION:
Early adolescence (10-13 years) is characterized by hormonal changes and accelerated physiological growth. Significant risk factors for the physical and mental health of children and adolescents include, among others, harmful physical activity, self-esteem and low self-esteem, and negative body image.

"Milli - a special shield for daily resilience" is a preventive intervention program. The main goal of the program is to raise adolescents' self-confidence and prevent negative self-image and body image as well as develop media literacy. In this study, the researchers will focus on the "Young Millie" program, designed for ages 10-12, fifth and sixth grades, and its core is the development of self-care. To increase the impact of the program on adolescents, the researchers developed a program that will be delivered to parents via a their adolescent children, as the 'agents of change'. Adloescents in the parent-component group will be given assignments to complete together with their parents at home, in coherence with the subject discussed in the weekly session of the school-based program.

The study will first evaluate the influence of parents on the program, and then evaluate the difference in adolescent outcomes from the program with or without this supplement.

Results will be measured using the study questionnaire, to be filled out by the adolescents before, after, and three months after the completion of the program. The questionnaire will include validated questionnaires with good psychometric qualities. Parents will fill out a satisfaction questionnaire before and after the program. The study protocol was approved by Tel Hai College institutional review board. Parents of all participants, in the intervention and in the control group, received information about the program and the study and were asked to provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of children 10-12 years old
2. 10-12-year-old children of participating parents
3. Participants who filled out the questionnaires before and after the program
4. Participants whose parents signed a letter of informed consent.

Exclusion Criteria:

1. Participants who didn't complete the questionnaires at baseline or at least twice.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Sociocultural Attitudes towards Appearance Questionnaire-4, Affects by Media subscale. | Measured three times over six months: at baseline, immediately after the program ends, and three months after the completion of the program, measuring a change in scores
  The Sociocultural Attitudes Towards Appearance Questionnaire (Schaefer et al., 2015). The investigators included the Media subscale, including 4 items. Items are rated on a 5-point scale: (1) always, (2) often, (3) sometimes, (4) rarely, (5) never. The total score is based on computing the average. A higher score indicates higher pressure from the media to change one's look.
Change from Baseline in Rosenberg Self Esteem Scale | Measured three times over six months: at baseline, immediately after the program ends, and three months after the completion of the program, measuring a change in scores
  Rosenberg Self Esteem Scale (Rosenberg, 1965)- 10 items. Scoring involves a method of combined ratings. Low self-esteem responses are "disagree" or
Change from Baseline in Body Esteem Scale | Measured three times over six months: at baseline, immediately after the program ends, and three months after the completion of the program, measuring a change in scores
  Body Esteem Scale- This questionnaire examines self-esteem of body and physical appearance and consists of 3 subscales: appearance (10 items), weight (8 items) and attribution 187 to others (5 items). Items are rated on a 5-point scale: (1) never, (2) rarely, (3) sometimes, (4) 188 often, and (5) always. A higher score indicates higher body-esteem (Mendelson, Mendelson, & White, 2001)
Change from Baseline in Advertising Scale | Measured three times over six months: at baseline, immediately after the program ends, and three months after the completion of the program, measuring a change in scores
  The Advertising scale contains 1 item- Identification of strategies used by media. This question is reflected as a protective factor. It contains 8 different strategies which participants choose from: higher number of strategies identified indicate better media literacy. (Golan et al., 2013).
Change from Baseline in Self-Caring | Measured three times over six months: at baseline, immediately after the program ends, and three months after the completion of the program, measuring a change in scores
  Developed by Prof. Moria Golan and assessed in previous research. Includes 14 items which are rated on a 4-point scale: (1) never, (2) rarely, (3) sometimes, (4) always. Items are summed, and higher scores indicate higher self-care behaviors. This questionnaire was designed to assess self care behaviors in adolescents.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Hai College, Kiryat Shmona, Upper Galilee, Israel

IPD SHARING:
Plan to Share IPD: No